CLINICAL TRIAL: NCT07372222
Title: Effect of a Posterior Shoulder Pillow on Pain and Sleep Quality After Rotator Cuff Repair: A Prospective Cohort Study
Brief Title: Effect of a Posterior Shoulder Pillow on Pain and Sleep Quality After Rotator Cuff Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhenlong, Associate Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20250422
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Injuries; Postoperative Pain; Sleep Quality
Keywords: Pillows; Rotator Cuff Repair; Postoperative Pain; Sleep Quality; Randomized Controlled Trial
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Pillow Group (Experimental): Patients who receive the standardized use of the posterior shoulder pillow in addition to the conventional rehabilitation protocol.
  Interventions: Device: Posterior Shoulder Pillow; Other: Conventional Rehabilitation Protocol
- Conventional Rehabilitation Group (Active Comparator): Patients who receive the conventional rehabilitation protocol only, without standardized use of the pillow.
  Interventions: Other: Conventional Rehabilitation Protocol

INTERVENTIONS:
Device: Posterior Shoulder Pillow — This is a standardized protocol for using a regular hospital ward pillow placed behind the shoulder (between the scapula and the bed) after arthroscopic rotator cuff repair. Patients in the intervention group are instructed to start using the pillow within 24 hours after surgery and maintain its use during rest and sleep for the 6-week study period. The pillow aims to provide support and improve comfort.
  Arms: Posterior Pillow Group
Other: Conventional Rehabilitation Protocol — This is the standard post-operative care for patients undergoing arthroscopic rotator cuff repair. It includes cryotherapy (ice packs), pharmacological analgesia (pain medication), and a progressive program of functional exercises guided by a physical therapist. This protocol is administered to all patients in the study, regardless of group assignment.

SUMMARY:
The goal of this clinical study is to learn if using a special pillow placed behind the shoulder can help to reduce pain and improve sleep for patients after surgery to repair a torn rotator cuff. The main questions it aims to answer are:

* Do patients who choose to use the posterior shoulder pillow have lower pain levels after surgery?
* Do these patients report better sleep quality during recovery?
* How safe and comfortable is the pillow for patients to use? Researchers will compare patients who use the pillow to those who do not use it to see if there is a difference in their recovery.

Participants will:

* Be asked about their willingness to use the pillow. Their treatment and recovery plan will be decided together with their doctor.
* Be asked to rate their pain and sleep quality several times after surgery: at 1 week, 2 weeks, 4 weeks, and 6 weeks.
* Have their shoulder function assessed by a clinician at 2, 4, and 6 weeks after surgery.
* Receive a standard MRI scan before and 6 weeks after surgery as part of their regular medical care to check on healing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rotator cuff tear, confirmed by imaging (MRI or ultrasound), and deemed suitable for either single-row or double-row arthroscopic repair surgery.
* Age between 40 and 70 years.
* Willing and able to provide written informed consent to participate in the study.
* Demonstrates good compliance with postoperative rehabilitation and follow-up requirements.

Exclusion Criteria:

* Presence of concomitant shoulder pathologies, such as glenohumeral osteoarthritis, adhesive capsulitis, history of labral repair, or irreparable tendon tears.
* Pre-existing severe shoulder infection, tumor, or other conditions that may significantly impact postoperative recovery.
* Previous history of shoulder surgery or severe shoulder deformity that could confound the assessment of postoperative outcomes.
* Cognitive impairment or inability to understand the pain assessment tools (e.g., VAS score).
* Significant comorbidities affecting the heart, liver, or kidneys, or requiring long-term use of medications that affect coagulation (e.g., aspirin).
* Diagnosis of malignant tumors or rheumatic autoimmune diseases that may interfere with postoperative recovery.
* MRI findings indicating significant fatty infiltration (>50%) or tendon retraction, suggesting potential compromise in surgical outcome and recovery.
* Superior migration of the humeral head or obliteration of the coracoacromial space, indicating a high difficulty of rotator cuff repair.
* Contraindications to postoperative rehabilitation exercises, such as severe osteoporosis or neuromuscular diseases.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain Score Measured by Visual Analog Scale (VAS) | From pre-operation (baseline) to 6 weeks post-operation.
  The Visual Analog Scale (VAS) for pain is a 100-mm horizontal line where 0 mm represents "no pain" and 100 mm represents "the worst pain imaginable." Higher scores indicate worse pain.
Sleep Quality Measured by the Pittsburgh Sleep Quality Index (PSQI) | From pre-operation (baseline) to 6 weeks post-operation.
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month interval. The global PSQI score ranges from 0 to 21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Shoulder Function | From pre-operation (baseline) to 6 weeks post-operation. Measured at 2 weeks, 4 weeks, and 6 weeks post-operation.
  Assessed by the Constant-Murley Score (CMS). The score ranges from 0 to 100, assessing pain, activities of daily living, range of motion, and strength, with higher scores indicating better function.
Tendon Healing Status Assessed by the Sugaya Classification on MRI | Measured at pre-operation (baseline) and at 6 weeks post-operation.
  Tendon integrity and healing will be evaluated on MRI using the Sugaya classification system. This is a 5-point scale (Type I-V) based on signal intensity and thickness of the repaired tendon, where Type I represents a fully healed tendon with sufficient thickness and low signal intensity, and Type V represents a re-tear. Lower grades indicate better tendon healing.
Muscle Fatty Infiltration Assessed by the Goutallier Classification on MRI | Measured at pre-operation (baseline) and at 6 weeks post-operation.
  The degree of fatty infiltration of the supraspinatus muscle will be evaluated on MRI using the Goutallier classification system. This is a 5-stage scale (Grade 0-4), where Grade 0 represents no fatty infiltration and Grade 4 represents >80% fatty infiltration. Higher grades indicate worse fatty degeneration.
Incidence of Complications | From immediately after intervention initiation up to 6 weeks post-operation. Assessed at each follow-up visit (24 hours, 1 week, 2 weeks, 4 weeks, 6 weeks).
  The occurrence of any adverse events related to the pillow use or rehabilitation, such as skin pressure ulcers, discomfort caused by the pillow, infection, etc.

OTHER OUTCOMES:
Subgroup Analysis of Intervention Effects | Assessed at the end of the study (after 6-week data collection).
  To explore the consistency of the intervention effect across different subgroups, as pre-specified in the study protocol. Subgroups are defined by:
  * Surgical technique (single-row vs. double-row suture repair)
  * Tear size/grade of rotator cuff tear

IPD SHARING:
Plan to Share IPD: No